CLINICAL TRIAL: NCT01742468
Title: Intervention With Products Enriched With Long Chain n-3 Polyunsaturated Fatty Acids (n-3 LC-PUFA) From Microalgae Oil in Patients With Rheumatoid Arthritis - Influence on Disease Activity and Inflammation Status
Brief Title: Intervention With Long-chain n-3 Polyunsaturated Fatty Acids From Microalgae Oil in Patients With Rheumatoid Arthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jena (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government)
Responsible Party: Principal Investigator, Gerhard Jahreis, Professor, University of Jena
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: H53-12
Record Dates: First submitted 2012-12-03; First posted 2012-12-05 (Estimated); Last update posted 2015-10-07 (Estimated); Status verified 2013-10

CONDITIONS: Rheumatoid Arthritis
Keywords: n-3 LC-PUFA, DHA, rheumatoid arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Sunflower Oil

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dietary supplement: n-3 LC-PUFA (Experimental): Name: microalgae oil (Schizochytrium sp., Maris DHA oil, no. 3790, IOI, Hamburg, Germany; rich in docosahexaenoic acid (DHA); Dosage: 8 g oil per day = 2.11 g DHA per day; Dosage form: 8g oil was included in 60 g sausage, 8 g tomato spread, 30 g milk powder
  Interventions: Dietary Supplement: long-chain n-3 PUFA
- Dietary supplement: sunflower oil (Placebo Comparator): Name: sunflower oil (PPM, Magdeburg, Germany); Dosage: 8 g per day; Dosage form: 8g oil was included in 60 g sausage, 8 g tomato spread, 30 g milk powder
  Interventions: Dietary Supplement: sunflower oil

INTERVENTIONS:
Dietary Supplement: long-chain n-3 PUFA — Dietary supplement: n-3 LC-PUFA = Microalgae oil (Schizochytrium sp., Maris DHA oil, no. 3790, IOI, Hamburg, Germany (rich in docosahexaenoic acid (DHA)); Dosage: 8 g oil per day = 2.11 g DHA per day; Dosage form: included in 60 g sausage, 8 g tomato spread, 30 g milk powder
  Other Names: n-3 LC-PUFA
  Arms: Dietary supplement: n-3 LC-PUFA
Dietary Supplement: sunflower oil — Dietary supplement: sunflower oil Name: sunflower oil (PPM, Magdeburg, Germany); Dosage: 8 g per day; Dosage form: 8g oil was included in 60 g sausage, 8 g tomato spread, 30 g milk powder
  Other Names: placebo
  Arms: Dietary supplement: sunflower oil

SUMMARY:
The study was performed to investigate the effects of a daily consumption of n-3 LC-PUFA supplemented products (sausage, tomato spread, milk beverage) on disease activity, inflammatory markers, and cardiovascular risk factors in patients with rheumatoid arthritis.

DETAILED DESCRIPTION:
Recent studies suggest that the daily intake of n-3 LC-PUFA (eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA)) can support the therapy of chronic-inflammatory diseases and might be useful to prevent coronary heart diseases. The majority of these studies do not differentiate between the effects of EPA and DHA. The present study investigate the therapeutic potential of DHA in patients with rheumatoid arthritis.

As a precondition for participating in this study, the patients were provided information in writing and verbally form about the details of the study. Written informed consent was obtained from all volunteers. Before the beginning of the study, all patients were subject to a medical examination by their general rheumatologist. Thirty-eight patients with rheumatoid arthritis (DAS ≥ 2.4) entered the study.

The placebo-controlled, randomized double-blind cross-over study consists of two investigation periods of 10 weeks, with a ten-week washout period in between (after the washout period the intervention was crossed between the groups and the respective products were consumed for further 10 weeks).

Patients in the placebo period receive 60 g sausage, 8 g tomato spread and 30 g milk powder (= 200 mL milk beverage) daily. These products were enriched with sunflower oil (8 g/d).

In the intervention period, the products (60 g sausage, 8 g tomato spread and 30 g milk powder (= 200 mL milk beverage) were enriched with 8 g microalgae oil (Schizochytrium sp., Maris DHA oil, no. 3790, IOI, Hamburg, Germany). In this group, the daily dose of docosahexaenoic acid (DHA) amounted to 2.11 g.

Venous blood is collected at the beginning and at the end of each period.

• Disease activity was determined by sum of tender and swollen joints (68/66), joint score DAS28, ultrasound score (US-7 score), rheumascan, inflammatory markers (ESR, C reactive protein), HAQ questionnaire and further lifestyle forms

ELIGIBILITY:
Inclusion Criteria:

* Patient has a diagnosis of RA (according to the ACR classification criteria, revised 2010) for at least 6 months prior to randomization.
* Patient has a moderate disease activity as defined by disease activity score DAS28 ≥ 2.4
* Patient has the ability to comprehend the full nature and purpose of the study, including possible risks and side effects, to cooperate with the investigator, to understand verbal and written instructions, and to comply with the requirements of the entire study.
* stable dosis of disease-modifying antirheumatic drugs within 4 weeks prior to randomization and presumably over the study periods (30 weeks).

Exclusion Criteria:

* Intra-articular corticosteroids within 4 weeks prior to randomization or blood sample taking
* Patients are permitted to receive either oral or parenteral glucocorticoids equivalent to ≤10 mg daily prednisone and nonsteroidal anti-inflammatory drug, if they have received a stable dose for at least 4 weeks prior to randomization and presumably over the study periods (30 weeks).

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2013-02; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Sum of tender and swollen joints (68/66), disease activity score DAS 28, ultrasound score US-7 | 10 weeks
  Disease activity parameters

SECONDARY OUTCOMES:
Inflammation markers such as erythrocyte sedimation rate (ESR), C reactive protein (CRP), adhesion molecules, cytokines, rheumascan | 10 weeks
  Further disease acitvity parameters
Concentrations of arachidonic acid, eicosapentaenoic acid, docosahexaenoic acid in plasma lipids and erythrocyte lipids | 10 weeks
  Precursors of eicosanoids (leukotriens, prostaglandins, thromboxanes) and docosanoids (resolvines)
Lipid mediators formed by lipoxygenases, cyclogenases | 10 weeks
  Lipidmediators derived from arachidonic acid, eicosapentaenoic acid, docosahexaenoic acid

OTHER OUTCOMES:
Blood lipids (total cholesterol, high density lipoprotein (HDL), low density lipoprotein (LDL), triacylglycerol (TAG), ox LDL, lipoprotein a) | 10 weeks
  Cardiovascular risk factors

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Jahreis, Professor, Principal Investigator — Friedrich Schiller University Jena, Department of Nutritional Physiology
Locations (2):
- Germany (2):
  - Facility: University of Jena, Institute of Nutrition, Department of Nutritional Physiology, Jena, Thuringia
  - Friedrich Schiller University, Clinic for Internal Medicine, Jena

REFERENCES:
- [Derived] Dawczynski C, Dittrich M, Neumann T, Goetze K, Welzel A, Oelzner P, Volker S, Schaible AM, Troisi F, Thomas L, Pace S, Koeberle A, Werz O, Schlattmann P, Lorkowski S, Jahreis G. Docosahexaenoic acid in the treatment of rheumatoid arthritis: A double-blind, placebo-controlled, randomized cross-over study with microalgae vs. sunflower oil. Clin Nutr. 2018 Apr;37(2):494-504. doi: 10.1016/j.clnu.2017.02.021. Epub 2017 Mar 6. PMID 28302406